CLINICAL TRIAL: NCT03032861
Title: Influence of the Prebiotic Effect of Orange Juice on the Bioavailability of Flavanones After Chronic Intake of Orange Juice.
Brief Title: The Prebiotic Effect of Daily Intake of Orange Juice Affects the Bioavailability of Flavanones?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Responsible Party: Principal Investigator, Thais Cesar, PhD, São Paulo State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SaoPSU2
Record Dates: First submitted 2017-01-06; First posted 2017-01-26 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Intestinal Diseases
Keywords: Orange juice; Microbiota; Prebiotic; Flavanones; Bioavailability
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Orange juice (Experimental): Ten women will consume 100% orange juice (300 mL/day) during 60 days.
  Interventions: Other: Orange juice

INTERVENTIONS:
Other: Orange juice — Thirty days before the beginning of trial, women (n= 10; BMI 23.8 kg/m2; 28 years) will be advised to not consumed foods containing prebiotic, probiotic and fibers, and citrus fruits and beverages. After 30 days, the participants will consume 300 mL of orange juice daily during 60 days. After 60 days of orange juice intervention, the participants will be submitted to 30 days of washout. Samples of blood, urine and feces will collect in five different occasions (baseline, 30 day, 60 day, 90 day, and 120 day) in order to evaluate the prebiotic effect of orange juice on gut microbiota and the bioavailability of its flavanones in blood, urine and feces.

SUMMARY:
This study aimed investigate the chronic effect of orange juice consumption on gut microbiota and in the bioavailability of flavanones and metabolites by feces, blood and urine analysis.

DETAILED DESCRIPTION:
Non-randomized study with interrupted time series and open-label, in which women were enrolled and advised to not consumed foods containing prebiotic, probiotic and fibers, and citrus fruits and beverages during 30 days before of intervention (n=10; BMI 23.8 kg/m2; 28 years). After 30 days, the participants will consume during 60 days 300 mL of orange juice daily. After 60 days of orange juice intervention, the participants will be submitted to 30 days of washout. Samples of blood, urine and feces will collect in five different occasions (baseline, 30 day, 60 day, 90 day, and 120 day) in order to evaluate the prebiotic effect of orange juice on gut microbiota and in the bioavailability of its flavanones. The recruitment process began in September 2016 and the intervention was carried out from October 2016 to February 2017, and the data analysis will start in February 2017. The sample number took into account variances on blood hesperitin levels with a type I error α = 0.05 and a type II error β = 0.2 (80% power) (Silveira et al., 2015). The minimum sample size should have six individuals into the same group. Considering an approximately 15% dropout rate, the final sample size of study was constituted by 10 women. Primary endpoint is the changes in total bacteria population (Lactobacillus spp., Bifidobacterium spp., and reduction of Clostridium spp.) that can result in increased of butyric, acetic, and propionic acid concentrations, and reduction of ammonium production. Secondary endpoint is enhancement of bioavailability of flavanones (hesperitin, naringenin) and metabolites in the blood, urine and feces. Kolmogorov Smirnov and Levene test will be used to assess the normality and homogeneity of data, respectively. One-way analysis of variance (ANOVA) will be apply to determine the intervention effect over the time 0, 30 day, 60 day, 90 day, and 120 day). P significance was set up ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

Healthy women BMI 18.5 - 29.9 kg/m2.

Exclusion Criteria:

Gastrointestinal diseases Pregnant women Regular use of medications Dietary restrictions, vegetarian diet, macrobiotic, etc. Use of vitamins or dietary supplements Use of probiotics or prebiotics in the last 3 months and antibiotics in the last 6 months.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Total counting of aerobic bacteria and facultative anaerobic bacteria | 4 months
Determination of butyric acid | 4 months
Determination of acetic acid | 4 months
Ammonium concentration | 4 mounths

SECONDARY OUTCOMES:
Bioavailability of hesperitin and naringenin in the blood, urine and feces | 4 months
  Quantification of hesperidin and naringenin and identification and quantification of their metabolites in the blood, urine and feces
Body mass index | 4 months
Body lean mass | 4 months
Body fat mass | 4 months
% body fat | 4 months
Ratio waist/hip | 4 mounths
Glucose | 4 mounths
Insulin | 4 mounths
Total cholesterol | 4 mounths
Low density lipoprotein cholesterol | 4 mounths
High density lipoprotein cholesterol | 4 mounths
Triglycerides | 4 mounths
hsCRP | 4 mounths
Alkaline phosphatase | 4 mounths
Aspartate enzyme aminotransferase | 4 mounths
Alanine enzyme aminotransferase | 4 mounths
GammaGT | 4 mounths
Glycemic curve | 4 mounths
Insulin curve | 4 mounths

CONTACTS AND LOCATIONS:
Overall Officials: Thais B Cesar, PhD, Principal Investigator — São Paulo State University
Locations (1):
- Sao Paulo State University "Julio de Mesquita Filho", Faculdade de Ciências Farmacêuticas, Araraquara, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
There is still no decision regarding if the individual participant data (IPD) will be available to other researchers.

REFERENCES:
- [Result] Silveira JQ, Cesar TB, Manthey JA, Baldwin EA, Bai J, Raithore S. Pharmacokinetics of flavanone glycosides after ingestion of single doses of fresh-squeezed orange juice versus commercially processed orange juice in healthy humans. J Agric Food Chem. 2014 Dec 31;62(52):12576-84. doi: 10.1021/jf5038163. Epub 2014 Dec 15. PMID 25495754
- [Result] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Result] Kanaze FI, Bounartzi MI, Georgarakis M, Niopas I. Pharmacokinetics of the citrus flavanone aglycones hesperetin and naringenin after single oral administration in human subjects. Eur J Clin Nutr. 2007 Apr;61(4):472-7. doi: 10.1038/sj.ejcn.1602543. Epub 2006 Oct 18. PMID 17047689